CLINICAL TRIAL: NCT02897648
Title: Evaluation of Pharmacokinetic / Pharmacodynamic and Tolerance Assessment of Dermal Administration of Beta-lactams in the Elderly
Acronym: BETALACUTANE
Status: Terminated | Type: Observational
Why Stopped: PI's decision
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: BETALACUTANE
Record Dates: First submitted 2016-09-01; First posted 2016-09-13 (Estimated); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Beta-Lactams; Aged Subject

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Assessment of dermal administration of Beta-Lactams — Evaluation of Pharmacokinetic / Pharmacodynamic of dermal administration of Beta-Lactams

SUMMARY:
The route of subcutaneous administration of drugs has become a common practice in some specialties (palliative care, geriatrics).

This is an alternative to oral, sublingual, rectal or intravenous Many drugs are used by subcutaneous route but few clinical studies evaluating the level of scientific relevance justifies their use.

The purpose of this study is to assess:

1. / Determine that there is no difference between the subcutaneously compared to intravenous administration in terms of dosage and serum PK / PD of Beta lactam objectives in a geriatric population.
2. / The safety and lack of toxicity of administrations subcutaneously.

Advantages disadvantages

* easy Of establishment
* Simplicity Monitoring and manipulation
* Reduced Risk of infection
* No Risk of venous thrombosis
* Lower cost Simple -Technique for support at home taking
* Limitation Aggressive gestures
* multiplicity Of all possible injection sites
* Technique Of choice for agitated patients or confused -Risk of localized edema (<1000mL / 24 / site)
* Use Impossible for some drugs
* Risk Discomfort and intolerance at the injection site

A practical study was conducted among 382 physicians (289 geriatricians and 93 infectious disease specialists). Among them 97.5% reported regular use of the subcutaneous route for the administration of antibiotics.

Declarative criteria pretend curb the use of this route was the lack of data Pk / Pd (61.2%); the absence of marketing authorization for the subcutaneous route (34.5%); the absence of serum assay available (2.1%).

DETAILED DESCRIPTION:
PROTOCOL

Primary objective :

• Determine that there is no difference between the subcutaneously compared to intravenous administration in terms of dosage and serum PK / PD objectives Beta lactam in a geriatric population.

Secondary objectives:

* Clinical evaluation at J14 and J90 (healing, death)
* Clinical tolerance of subcutaneously by self-assessment or hetero-evaluation of the existence of cognitive disorders

Monitoring of antibiotic dosages:

* Making systematic assay serum concentrations of residual antibiotics in the range of 30 min prior to reinjection H24 after starting treatment and then weekly monitoring.
* Realization of the assays according to the method of Liquid Chromatography-Mass Spectrometry (LC-MS)

Patient monitoring of J1-J14:

• Clinical monitoring and biological usual

ELIGIBILITY:
Inclusion Criteria:

* Geriatric Population (≥ 75 years)
* Infection may cause bacteremia or not: Gram-negative bacilli and gram-positive cocci susceptible to beta-lactam

Exclusion Criteria:

* Patient Refusal expressed or legal guardian
* polymicrobial infection

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged of >74 years old with Gram-negative bacilli and gram-positive cocci susceptible to beta-lactam
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2015-06-26 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2023-03-06 (Actual)

PRIMARY OUTCOMES:
Assessment of change of residual concentration of Beta-Lactam antibiotic | Minute 30, hour 24, Day 7. Then once a Week 2, 3, 4, 5, 6, 7, 8, 9, 10, 11 and 12
  • Making systematic assay serum concentrations of residual antibiotics in the range of 30 min prior to reinjection H24 after starting treatment and then weekly monitoring.an

SECONDARY OUTCOMES:
Assessment of patient healing (infection free) | Day 14 and day 90
  Evaluation of healing to day 14 and day 90. The answer should be: Yes / No

CONTACTS AND LOCATIONS:
Overall Officials: EL HELALI Najoua, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided